CLINICAL TRIAL: NCT07244796
Title: Developing Healthy Lifestyle Behaviors in High School Students: An Experimental Education Model
Brief Title: Promoting Healthy Lifestyle Behaviors in High School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ErzrurumTU
Record Dates: First submitted 2025-09-09; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy Lifestyle Behaviors in High School Students
Keywords: Adolescents; Healthy lifestyle behaviors; Hygiene; Screen dependency; Physical activity; Nutrition; Sleep habits; Health-related quality of life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental pretest-posttest design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group trained (Experimental): During the research process, training was provided on Hygiene, Screen addiction, Physical activity, Nutrition and Sleep habits to encourage healthy living behaviors.
  Interventions: Behavioral: provide training
- Control group (Active Comparator): After the research process was completed and the pretest and posttest data were collected, training was provided on Hygiene, Screen addiction, Physical activity, Nutrition and Sleep habits to encourage healthy living behaviors.
  Interventions: Behavioral: provide training

INTERVENTIONS:
Behavioral: provide training — Face-to-face training on hygiene practices, screen addiction, nutrition, physical activity, and sleep habits

SUMMARY:
Adolescence (ages 10-19) is a critical developmental stage in which individuals undergo significant physical, psychological, and social changes. Health behaviors acquired during this period often persist into adulthood, directly influencing both individual and public health. Adolescents' lifestyles are shaped by factors such as family, school, peers, and socio-cultural environment. A healthy lifestyle includes habits such as regular physical activity, balanced nutrition, adequate sleep, and limited screen time, all of which are key determinants of quality of life.

The aim of this study is to evaluate the effectiveness of an educational program designed to improve high school students' hygiene, screen use, nutrition, physical activity, and sleep habits. It is hypothesized that the program will increase students' healthy lifestyle beliefs and hygiene behaviors, while reducing screen addiction and insomnia levels.

DETAILED DESCRIPTION:
Adolescence, defined by the World Health Organization as the period between 10 and 19 years of age, represents a transitional stage from childhood to adulthood characterized by profound physiological, cognitive, psychological, and social changes. These transformations significantly influence adolescents' health-related quality of life, which is a multidimensional construct encompassing physical, psychological, and social well-being. Health behaviors acquired during this developmental stage tend to persist into adulthood and therefore play a critical role in the prevention of chronic diseases and the promotion of lifelong health. For instance, unhealthy dietary patterns, sedentary lifestyles, excessive screen use, and irregular sleep habits established during adolescence may increase the risk of obesity, cardiometabolic disorders, and psychological problems in later life. Conversely, adopting positive health practices such as balanced nutrition, regular physical activity, proper sleep hygiene, and limited screen time during this period can enhance quality of life and support healthy growth and development.

Adolescents' health behaviors are influenced by multiple environmental factors, including family, peers, school, socioeconomic status, and cultural context. Thus, interventions aimed at promoting healthy lifestyles in this age group require a holistic and multifactorial approach. Education programs focusing on health-related knowledge and practices have been shown to play a key role in shaping positive behaviors and raising awareness about health protection and disease prevention.

The present study aims to evaluate the effectiveness of an educational program designed for high school students, addressing five key domains: hygiene, screen dependency, nutrition, physical activity, and sleep habits. The program seeks not only to increase adolescents' knowledge in these areas but also to instill sustainable health-promoting behaviors. Four hypotheses were established: (1) students in the intervention group will report higher scores on the Healthy Lifestyle Beliefs Scale compared to the control group; (2) their Screen Dependency Scale scores will decrease; (3) their Hygiene Behaviors Scale scores will increase; and (4) their Bergen Insomnia Scale scores will decrease following the program.

This research emphasizes the importance of implementing structured, school-based educational interventions to promote healthier lifestyles among adolescents. By targeting multiple dimensions of health simultaneously, such interventions may contribute to reducing long-term health risks, improving well-being, and fostering healthier future generations.

ELIGIBILITY:
Inclusion Criteria:

* Being a 9th, 10th, or 11th grade student
* Having no illness that may cause communication problems
* Willingness to participate in the study

Exclusion Criteria:

* Being a 12th grade student
* Having any illness that prevents communication
* Unwillingness to participate in the study

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Healthy Lifestyle Belief Scale for Adolescents | Week 1 = Data collection from all participants. Weeks 2, 3, 4, 5, and 6 = Training provided to the Training Group. Week 7 = Post-test data collection from all participants. Weeks 8, 9, 10, 11, and 12 = Training provided to the Control Group.
  The Healthy Lifestyle Belief Scale for Adolescents was developed by Kelly et al. (2011), and its Turkish validity and reliability study was conducted by Kudubeş and Bektas (2020). The scale highlights beliefs related to various aspects of maintaining a healthy lifestyle. The scale has a total of 16 items and three subscales.The scale, prepared according to a five-point Likert system, is answered on a scale of "1 = Strongly Disagree" to "5 = Strongly Agree." A minimum of 16 and a maximum of 80 points can be obtained on the entire scale. An increase in the score obtained on the scale indicates an increase in adolescents' belief in healthy living. The Cronbach's alpha coefficient of the scale is 0.90.
Screen Addiction Scale | Week 1 = Data collection from all participants. Weeks 2, 3, 4, 5, and 6 = Training provided to the Training Group. Week 7 = Post-test data collection from all participants. Weeks 8, 9, 10, 11, and 12 = Training provided to the Control Group.
  The SAS is a comprehensive measurement tool that covers any screen rather than focusing on specific screen-based devices. The scale can be defined as a synthesis of screen-based addictions such as internet, smartphone, television, social media, computer, and video game addiction. It has been found that the EBÖ has a structure consisting of 21 items and 4 factors. A valid and reliable scale was obtained, validated by a first-order multifactor model and a second-order multifactor model. The scale, prepared according to a five-point Likert system, is answered as "1=Strongly Disagree, 5=Strongly Agree." The scale can yield a minimum score of 21 and a maximum score of 105. High scores on the scale indicate high screen dependency, while low scores indicate low screen dependency. The Cronbach's alpha value, which is the internal consistency coefficient of the scale, is reported to be 0.925.

SECONDARY OUTCOMES:
Hygiene Behavior Assessment Scale | 4 Week 1 = Data collection from all participants. Weeks 2, 3, 4, 5, and 6 = Training provided to the Training Group. Week 7 = Post-test data collection from all participants. Weeks 8, 9, 10, 11, and 12 = Training provided to the Control Group.
  The HBAS, developed by Gül and Özay Köse (2020), has been reported to be a valid and reliable measurement tool for assessing hygiene behaviors among secondary school students. The HBAS consists of a total of 27 items, all prepared on a 5-point Likert scale, and comprises two factors. The statements in the scale are scored using the following scale: 1: Never, 2: Rarely, 3: Sometimes, 4: Very often, 5: Always. Thus, the lowest possible score on the HDÖ is 27, and the highest possible score is 135. The Cronbach Alpha internal consistency coefficient for the scale as a whole is reported as .902.
Bergen Insomnia Scale (BIS) in Adolescents | Week 1 = Data collection from all participants. Weeks 2, 3, 4, 5, and 6 = Training provided to the Training Group. Week 7 = Post-test data collection from all participants. Weeks 8, 9, 10, 11, and 12 = Training provided to the Control Group.
  The scale developed by Pallesen et al. (2008) was validated and tested for reliability in Turkish by Bay and Ergun (2018). The Bergen Insomnia Scale reliability and validity study indicated that it can be used to measure insomnia in adolescents in Turkish society. The scale consists of six questions with two factors. The scale, which tests different symptoms of insomnia, is an 8-point Likert scale. The lowest possible score on the scale is 0, and the highest possible score is 42. Within the scope of reliability analyses, it was stated that the Cronbach's alpha reliability coefficient of the scale was 0.79 for the daytime symptoms subscale, 0.63 for the nighttime symptoms subscale, and 0.72 for the total BIS

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No